CLINICAL TRIAL: NCT01533220
Title: A Randomized, Double-blind, Prospective, Multicentric, Superior Efficacy and Safety of Naphazoline Hydrocloride + Pheniramine Maleate + Panthenol Compared With Naphazoline Hydrocloride in the Symptomatic Control of Nasal Congestion and Nasopharyngeal Due to Colds or Other Upper Respiratory Allergies
Brief Title: Efficacy of Nasal Naphazoline Hydrocloride + Pheniramine Maleate + Panthenol Compared With Naphazoline Hydrocloride in the Symptomatic Control of Nasal Congestion and Nasopharyngeal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMPEMS1011
Record Dates: First submitted 2012-02-09; First posted 2012-02-15 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Flu; Cold; Allergic Disorder of Respiratory System
Keywords: nasal and nasopharyngeal congestion
MeSH Terms: conditions — Influenza, Human; Common Cold | interventions — Pheniramine; dexpanthenol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Naphazoline Hydrocloride (1.0mg) + Pheniramine Maleate (0.2mg) + Panthenol(5.0mg).
  02 drops in each nostril every 12 hours for 3 days
  Interventions: Drug: Naphazoline hydrocloride + Pheniramine Maleate + Panthenol
- Comparator group (Active Comparator): Naphazoline Hydrocloride (0.5mg)
  02 drops in each nostril every 12 hours for 3 days
  Interventions: Drug: naphazoline hydrocloride

INTERVENTIONS:
Drug: naphazoline hydrocloride — 02 drops into each nostril, 04 times a day for 03 days
  Arms: Comparator group
Drug: Naphazoline hydrocloride + Pheniramine Maleate + Panthenol — 02 drops into each nostril each 12 hours for 03 days
  Arms: Test group

SUMMARY:
The common cold is a major cause of nasal obstruction and reaches children and adults two or more times a year. At the moment, there is no cure for the common cold, and therefore the reduction of symptoms is the focus of the treatment.

The study has parallel distribution design, with two equal groups, in which one group will be treated by a combination of naphazoline hydrocloride + pheniramine maleate + panthenol and the other will receive treatment with naphazoline hydrocloride.

DETAILED DESCRIPTION:
STUDY DESIGN

* randomized,double blind, prospective, multicentric, parallel group, intent to treat trial
* Experiment duration: 3 days
* 2 visits (days 0 and 2)
* Evaluation of symptoms reduction
* Adverse events evaluation

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to understand the study procedures, agree to participate and give written consent.
2. Patients aged over 18 years of both sexes;
3. Patients with clinical signs of flu and colds or other upper respiratory allergies;
4. Patients with early signs and symptoms with time of evolution not more than 72 hours.

Exclusion Criteria:

1. Patients treated with antibiotics
2. Current treatment with immunosuppressants (eg.cyclosporine or methotrexate);
3. Use of intranasal cromalin the week before inclusion;
4. Use of decongestants or anti-histaminic (intranasal or systemic);
5. Presence of any disease or anatomical abnormality that may difficult the data analysis ;
6. Uncontrolled hypertension;
7. Presence of respiratory symptoms for more than 14 days;
8. History of abuse of drugs and alcohol;
9. Presence of other concomitant pulmonary diseases;
10. Hypersensitivity to any compound of investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2013-08-31 (Actual); Study Completion 2014-04-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment in nasal congestion reduction based on Peak Flow Nasal Inspiratory (PFNI) assay | 3 days
  The individual response rate to the nasal congestion reduction is calculated by measuring the peak flow nasal inspiratory (PFNI) during the first and last visit.

SECONDARY OUTCOMES:
Safety will be evaluated by the Adverse events occurence | 3 days
  Adverse events will be collected and followed in order to evaluate safety and tolerability